CLINICAL TRIAL: NCT07377058
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study on the Efficacy and Safety of Tocilizumab in the Treatment of Anti-MDA5 Antibody-Positive Adult Dermatomyositis
Brief Title: RCT of Tocilizumab for Anti-MDA5+DM
Acronym: PROMIS-MDA5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wang Qian, Prof, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I-25PJ1573
Record Dates: First submitted 2025-11-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — tocilizumab; Glucocorticoids; Tacrolimus; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCZ (Experimental)
  Interventions: Biological: Tocilizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Biological: Tocilizumab — Tocilizumab is a humanized monoclonal antibody targeting the IL-6 receptor, exerting therapeutic effects by specifically blocking the IL-6 signaling pathway.
  Other Names: Glucocorticoids; tacrolimus; ciclosporin
  Arms: TCZ
Drug: Standard medical treatment — Standard medical treatment for patients with anti-MDA5+ dermatomyositis
  Other Names: Glucocorticoids; tacrolimus; ciclosporin
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if tocilizumab works to treat anti-MDA5+ dermatomyositis (anti-MDA5+DM) in adults. It will also learn about the safety of tocilizumab. The main questions it aims to answer are:

Does tocilizumab improve patients' clinical symptoms? Does tocilizumab improve patients' respiratory failure? What medical problems do participants have when taking tocilizumab? Researchers will compare tocilizumab to a placebo (a look-alike substance that contains no drug) to see if tocilizumab works to treat patients with anti-MDA5+ DM.

Participants will:

Take tocilizumab or a placebo every two weeks for 2 months Visit the clinic once every 2 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria must be met for eligibility:

  1. Age ≥ 18 years and < 65 years; no gender restriction; total body weight ≥ 45 kg;
  2. Diagnostic Criteria for Anti-MDA5-DM: Refer to the "2023 Chinese Expert Consensus on Diagnosis and Treatment of Anti-Melanoma Differentiation-Related Gene 5 Antibody-Positive Dermatomyositis in China." Dermatomyositis patients exhibiting one of the following manifestations-Gottron's papules, Gottron's rash, or erythema ab igne-along with positive serum anti-MDA5 antibodies, may be diagnosed with anti-MDA5-DM;
  3. If patients have concomitant ILD, the following conditions must be met: i) Pulse oxygen saturation (SpO₂) ≥ 90% or PaO₂ ≥ 60 mmHg; ii) Pulmonary function tests showing forced vital capacity percentage of predicted (FVC%) ≥ 60% and carbon monoxide diffusion capacity percentage of predicted (DLco%) ≥ 40%; iii) High-resolution chest CT demonstrating pulmonary interstitial lesions involving < 50% of lung fields;
  4. Patients must have received oral prednisone (< 1 mg/kg/day, or equivalent dose of other glucocorticoids) for ≥ 4 weeks prior to randomization;
  5. Patients must have received a stable dose of a calcineurin inhibitor (CNI, such as cyclosporine or tacrolimus) for ≥4 weeks prior to randomization; if immunosuppressive therapy was discontinued prior to the screening visit, a washout period of at least 4 weeks is required;
  6. Patients must receive prophylactic treatment with trimethoprim-sulfamethoxazole (TMP-SMZ, 400mg trimethoprim/80mg sulfamethoxazole) 1-2 tablets daily during treatment;
  7. Women of childbearing potential must have a negative pregnancy test at study entry. If sexually active, they must agree to use effective contraception throughout the study period and must not intend to become pregnant during the study.
  8. Patients voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

* 1. Polymyositis, anti-synthetase syndrome, immune-mediated necrotizing myositis, or overlap myositis with other connective tissue diseases; 2. Patients with life-threatening complications, including but not limited to acute coronary syndrome (e.g., myocardial infarction, unstable angina) within 24 weeks prior to screening or any history of significant cerebrovascular disease; 3. Any of the following laboratory abnormalities at screening: white blood cell count <3.0×10⁹/L, neutrophil count <1.0×10⁹/L, lymphocyte count <0.5×10⁹/L, hemoglobin <90 g/L, platelet count <50×10⁹/L; severe hepatic impairment (ALT or AST ≥3 times ULN, total bilirubin ≥1.5 times ULN, excluding serum ALT or AST elevation due to dermatomyositis); severe renal impairment (creatinine clearance ≤45 mL/min); 4. Patients hospitalized for severe infection within 60 days prior to screening, or who received intravenous antibiotics (patients who used intravenous antibiotics must complete a five-half-life washout period and confirm absence of active infection before enrollment), but may receive empirical oral antibiotics or topical antibiotics; 5. Active tuberculosis infection that is untreated or inadequately treated; Latent tuberculosis infection (LTBI) requires at least 2 weeks of preventive antituberculosis therapy (including at least 2 antituberculosis drugs) prior to randomization, continuing through study completion. LTBI is defined as: Positive IGRA result (acceptable IGRA assays include: QFT-GIT, QFT-G, and T-spot® TB test); 6. Active viral hepatitis at screening: HBsAg-positive, HBeAg-positive, or HBV-DNA >10³ copies/L (HBV-DNA testing required if HBcAb-positive); HCVAb-positive; 7. Documented HIV infection, evidenced by positive serological test results or positive HIV serological test results at screening; 8. If the patient develops ILD-related clinical manifestations or progressive radiographic worsening within 4 weeks, RP-ILD should be considered. RP-ILD is defined as the presence of any one of the following four conditions within 1 month after the onset of respiratory symptoms: ① Acute and progressive worsening of dyspnea requiring hospitalization or supplemental oxygen; ② Decline in pulmonary function, manifested as a decrease in FVC% >10% with or without a decrease in DLco% >15%; ③ Increased interstitial abnormalities on chest HRCT scan >20%; ④ Decrease in arterial blood gas or partial pressure of oxygen >10 mmHg, indicating respiratory failure; and PaO₂/FiO₂≥200 mmHg.

  9. Allergy to the active ingredient tocilizumab or any of its excipients; 10. Patients with sulfonamide allergy; 11. Patients unable to complete pulmonary function testing at baseline; 12. Patients receiving prednisone at a dose exceeding 2 mg/kg/day prior to screening; 13. Patients receiving intravenous immunoglobulin (IVIG) prior to screening must discontinue treatment for at least 30 days; 14. Patients who used one or more of the following medications within the specified time window prior to screening:
  1. Rituximab within 6 months prior to screening;
  2. JAK inhibitors within 2 weeks prior to screening;
  3. Use of other biologics (including but not limited to anakinra, adalimumab, infliximab) or other immunosuppressive agents (including but not limited to methotrexate, azathioprine, mycophenolate mofetil) within 4 weeks prior to screening; 15. Patients with prior use of the study drug, other IL-6 inhibitors, or analogues; 16. Pregnant or lactating women, or women planning to become pregnant or initiate lactation; 17. History of malignant tumors within the past 5 years (excluding adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical carcinoma in situ with no evidence of recurrence within the preceding 5 years); 18. Other conditions deemed ineligible for study inclusion by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
TIS improvement | at Week 16 of treatment
  Proportion of patients achieving minimal improvement in Total Improvement Score (TIS≥20)
ILD improvement | at Week 16
  Change in PaO2/FiO2 ratio from baseline (patients with concomitant ILD)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT07377058/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT07377058/ICF_001.pdf